CLINICAL TRIAL: NCT01204736
Title: A Comparison of Two Surgical Procedures That Restore Elbow Extension
Brief Title: Comparing Outcomes of Elbow Extension Tendon Transfers
Status: Completed | Type: Observational
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Collaborators: Shirley Ryan AbilityLab (Other); Northwestern University (Other); Case Western Reserve University (Other); Loyola University (Other); MetroHealth System, Ohio (Other)
Responsible Party: Sponsor
Other Study IDs: B7515-R
Record Dates: First submitted 2010-09-15; First posted 2010-09-17 (Estimated); Results first posted 2016-01-07 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-02

CONDITIONS: Cervical Spinal Cord Injury
Keywords: tendon transfer; elbow

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Group 1: Subjects with posterior deltoid-to-triceps tendon transfers
- Group 2: Subjects with biceps-to-triceps tendon transfers
- Group 3: Subjects with cervical SCI who have not had tendon transfers
- Group 4: Unimpaired control subjects

SUMMARY:
Active elbow extension has significant functional benefits for individuals with tetraplegia. The proposed work will provide information to assess how effectively people are using their elbow extension tendon transfers, and whether one surgery works more effectively than the other. This study will provide recommendations to clinicians about the possibility of improving function after surgery using rehab techniques.

DETAILED DESCRIPTION:
Voluntary control of elbow extension significantly improves functional abilities for individuals with tetraplegia. As a result, surgical reconstruction of elbow extension via tendon transfer is considered a fundamental intervention that benefits the patient, even if other tendon transfers aimed at improving hand function are never performed. Presently, there are two common tendon transfer surgeries used to restore elbow extension following spinal cord injury. These are the posterior deltoid to triceps transfer and the biceps to triceps transfer. Both surgeries significantly improve voluntary elbow extension, although there is variability in the amount of control that is restored among patients. This study will directly compare the performance of the posterior deltoid transfer to the biceps transfer with regard to: voluntary elbow extension strength, the ability to activate the transfer, and neural factors associated with voluntary and involuntary control of individual muscles. These comparisons will be made in functionally relevant postures and will provide fundamental information that will improve clinical understanding of the capacity of each of these two procedures to restore elbow extension.

The fundamental hypothesis of this proposal is that an inability to maximally activate the transferred posterior deltoid and the transferred biceps significantly limits the elbow extension moment that can be produced.

ELIGIBILITY:
Inclusion Criteria:

* Cervical Spinal Cord Injury (C5-C7)
* Posterior Deltoid to Triceps Tendon Transfer at least one year post-surgery
* Biceps to Triceps Tendon Transfer at least one year post-surgery

Exclusion Criteria:

* Subjects will be excluded from the studies if there is presence of concurrent severe medical illness, including:

  * unhealed decubiti
  * use of baclofen pumps
  * existing infection
  * cardiovascular disease
  * significant osteoporosis (as indicated by a history of fractures following injury)
  * or a history of pulmonary complications or autonomic dysreflexia

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Three groups of subjects will be recruited to participate in the experiments: individuals that have had the posterior deltoid to triceps tendon transfer, individuals that have the biceps to triceps tendon transfer, and individuals with SCI between C5-C7 who have not had tendon transfers. Nominally, we plan to recruit 15 subjects from each group.
Sampling Method: Non-Probability Sample
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2014-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wendy M Murray, PhD, Principal Investigator — Edward Hines Jr. VA Hospital, Hines, IL
Locations (1):
- Edward Hines Jr. VA Hospital, Hines, IL, Hines, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Started | 4 | 5 | 3 | 2
Completed | 4 | 5 | 3 | 2
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4 | Total
Number analyzed (Participants) | 4 | 5 | 3 | 2 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.8 (7.3) | 26.6 (8.2) | 45.2 (11.5) | 33.5 (0.7) | 37.3 (12.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 0 | 1 | 3
  Male | 2 | 5 | 3 | 1 | 11

OUTCOME MEASURES:

1. Primary Outcome: Elbow Extension Strength
Description: Elbow extension strength was measured as the maximum elbow extension moment that subject's could generate. We used an elbow moment transducer to measure elbow moments under isometric (no change in arm posture) conditions. Subjects performed three trials at maximum effort, holding maximum elbow extension for 5 to 7 seconds. The maximum moment was computed as the maximum average moment sustained over a 0.5 second window.
Time Frame: At least one year post surgery
Measure: Mean (Standard Deviation); unit: Newton-Meters
Units Other Than Participants: Upper limbs
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Number analyzed (Participants) | 4 | 5 | 3 | 2
Number analyzed (Upper limbs) | 6 | 7 | 3 | 2
Newton-Meters | 2.74 (0.22) | 8.8 (3.9) | 0 (0) | 68.7 (12.3)

ADVERSE EVENTS:
Arm/Group | Group 1 | Group 2 | Group 3 | Group 4
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5 | 0/3 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No